CLINICAL TRIAL: NCT01585519
Title: Effect of Increased Whole Apple Consumption, Apple Extract and Freeze-dried Apple Products on Biomarkers of Cardiovascular Disease Risk: a Randomised Intervention in Participants at Increased Risk of Cardiovascular Disease
Brief Title: A Study Examining Effects of Apples/ Apple Products on Heart Disease Risk
Acronym: APPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Reader, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11.22v5
Record Dates: First submitted 2012-04-19; First posted 2012-04-26 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Disease
Keywords: High Epicatechin Apples; Low Epicatechin Apples; Apple Extract; Apple Granules; Blood Pressure; Cholesterol
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- (Group 1) Low Apple Diet (No Intervention)
- (Group 2) 2 High Apples (Experimental)
  Interventions: Dietary Supplement: High/ Low Epicatechin Apples/ Apple Extract/ Granules
- (Group 3) 2 Low Apples (Experimental)
  Interventions: Dietary Supplement: High/ Low Epicatechin Apples/ Apple Extract/ Granules
- (Group 4) 2 x 4.4g apple granules (Experimental)
  Interventions: Dietary Supplement: High/ Low Epicatechin Apples/ Apple Extract/ Granules
- (Group 5) 2 x Apple Extract Capsules (Experimental)
  Interventions: Dietary Supplement: High/ Low Epicatechin Apples/ Apple Extract/ Granules

INTERVENTIONS:
Dietary Supplement: High/ Low Epicatechin Apples/ Apple Extract/ Granules — (Group 1) Low Apple Diet (i.e. <1 portion per day) + 2 placebo capsules daily.
  (Group 2) 2 x High Epicatechin Apples daily + 2 placebo capsules daily.
  (Group 3) 2 x Low Epicatechin Apples daily + 2 placebo capsules daily.
  (Group 4) Low apple diet + 2 x 4.4g of apple granules daily + 2 placebo capsules daily.
  (Group 5) Low apple diet + 2 x Apple Extract Capsules daily.
  Other Names: High Polyphenol Apples; Low Polyphenol Apples
  Arms: (Group 2) 2 High Apples; (Group 3) 2 Low Apples; (Group 4) 2 x 4.4g apple granules; (Group 5) 2 x Apple Extract Capsules

SUMMARY:
This study will examine if health benefits of consuming nutrient-rich apples, an apple extract and freeze dried apple product will be similar. 50 volunteers at increased risk of heart disease will consume either a low apple diet (<1 portion/d), 2 high or low polyphenol apples/day, an apple extract, or freeze dried apple granule product for 4 weeks (ten participants per group, randomly assigned). Apart from the extract group, all volunteers will consume a placebo. All volunteers will follow a low apple diet (<1 apple per day) other than what has been provided by the research team. Volunteers will complete food diaries at the start and end of the study and a number of questionnaires. Blood and urine samples collected at 0 and 4 weeks

DETAILED DESCRIPTION:
Many products (such as bioactive extracts) attempt to replicate health benefits of a diet rich in fruit and vegetables, however, it is not known whether similar health benefits can be gained from consuming these processed products. A placebo-controlled intervention study will examine if health benefits are similar between products. Volunteers will have one risk factor for heart disease. Recruitment will be by advertisement from QUB and general public. Apples/apple products will be provided for the 4 weeks, but otherwise volunteers' normal diet and lifestyle will be followed. Blood and urine samples will be collected at week 0 and week 4. 4-day food diaries will be completed at the start and end of the study. A number of questionnaires (physical activity, lifestyle, levels of liking, tolerability to study products, study evaluation) will be completed at the start and end of the study. As this is a pilot study, power calculations were not considered appropriate. Statistical analysis will be carried out in SPSS, each endpoint of interest from the week 0 measure will be compared between the five intervention groups by one way analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* > 50 years old or
* Current Smoker or
* Systolic Blood Pressure 120-139mmHg/ Diastolic Blood Pressure 80-89mmHg or
* Total Cholesterol >5.2mmol/l or HDL cholesterol <1.03mmol/l or
* BMI >25 kg/m2

Exclusion Criteria:

* Diabetes mellitus
* An acute coronary syndrome or transient ischaemic attack within the past 3 months
* Special dietary requirements, food sensitivities or vegetarian/ vegan diet by choice
* Oral anticoagulation therapy
* BMI >35 kg/m2
* Excessive alcohol consumption (>28 U/week men or >21 U/week women)
* Pregnancy/ lactation
* Taking antioxidant supplements
* Medical conditions or dietary restrictions that would substantially limit ability to complete the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Between group change in oxidised-LDL | Weeks 0 and 4

SECONDARY OUTCOMES:
Between group change in self-reported apple or apple product intake | Weeks 0 and 4
Between group change in biochemical markers of nutritional status | Weeks 0 and 4
  Polyphenol levels (including epicatechin and quercetin) in plasma. Vitamin C and carotenoid concentrations in serum. Polyphenol and carotenoid concentrations in LDL.
Between group change in biomarkers of cardiovascular disease risk | Weeks 0 and 4
  Blood pressure will be measured twice from the right arm, using an automated Omron sphygmomanometer, with the participant sitting quietly for at least five minutes.
  Total cholesterol, HDL cholesterol and triglycerides in serum will be measured using automated enzymatic assays.
  High sensitivity CRP will be assessed by automated immunoassay.
  Weight will be monitored weekly over the 4 week intervention.
Between group change in other biomarkers of cardiovascular disease risk | Weeks 0 and 4
  Isoprostanes in urine by ELISA. Serum ICAM-1, VCAM-1 and E-selectin, LDL particle size, malondialdehyde in serum by HPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Jayne V Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (2):
- United Kingdom (2):
  - Queen's University Belfast, Belfast, Northern Ireland
  - Queen's Unversity, Belfast, Belfast, Northern Ireland